CLINICAL TRIAL: NCT04164732
Title: A Multi-center, Randomized, Placebo-controlled Patient and Investigator-blinded Study to Explore the Efficacy of Oral Sacubitril/Valsartan in Adult Patients With Non-obstructive Hypertrophic Cardiomyopathy (nHCM)
Brief Title: Study of Efficacy of Oral Sacubitril/Valsartan in Adult Patients With Non-obstructive Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696I12201; 2019-003098-24 (EudraCT Number)
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: non-obstructive; hypertrophic cardiomyopathy; genetic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigator and subject will be blinded to treatment allocation during the treatment period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LCZ696 BID (Experimental): Patients were treated with LCZ696. The target dose level was 200 mg p.o. b.i.d.
  Interventions: Drug: LCZ696
- Placebo BID (Placebo Comparator): Placebo to LCZ696
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — LCZ696 orally twice daily
  Other Names: sacubitril; valsartan
  Arms: LCZ696 BID
Drug: Placebo — placebo
  Arms: Placebo BID

SUMMARY:
The purpose of this study was to determine if LCZ696 can improve functional capacity (via improved peak VO2) in non-obstructive hypertrophic cardiomyopathy (HCM) patient population over the course of 50 weeks of treatment.

DETAILED DESCRIPTION:
This was a multi-center, placebo-controlled, patient and investigator-blinded study in non-obstructive HCM patients.

The study comprised a ≤ 35-day screening/baseline period, a 4-week single-blind treatment run-in period, followed by a 46-week double-blind placebo-controlled treatment period (total treatment period of 50 weeks), and a follow-up period approximately 30 days after the last dose.

The treatment run-in period was planned to ensure that as large a proportion as possible of patients:

1. had stable symptoms and could comply with study visits, and
2. could tolerate at least low dose LCZ696. During the run-in period, all patients received oral (p.o.) placebo b.i.d. for 2 weeks followed by 50 mg p.o. of active LCZ696 b.i.d. for 2 weeks. Patients who were unable to tolerate either placebo or the 50 mg p.o. b.i.d. dose level, were considered treatment run-in failures and were neither randomized into the double-blind, placebo-controlled study, nor included in the efficacy analysis.

In the double-blind treatment period, participants were randomized 1:1 to placebo or LCZ696. In the LCZ696 arm, participants started at a LCZ696 100 mg p.o. b.i.d dose. After approximately 14 days, patients who tolerated the 100 mg p.o. b.i.d. dose were up-titrated to 200 mg p.o. b.i.d. dose, whereas those who did not meet the safety criteria were titrated back down to the 50 mg b.i.d. dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hypertrophic Cardiomyopathy with a left ventricular wall thickness greater than or equal to 13mm as determined by the echocardiogram obtained during the screening/baseline period
* Left ventricular ejection fraction (LVEF) greater than or equal to 50% as determined by echocardiogram obtained during the screening/baseline period
* Symptoms consistent with New York Heart Association (NYHA) Class II-III heart failure by physician assessment, or asymptomatic/NYHA Class I patients with:

  * NT-proBNP blood sample levels above 250 pg/ml and
  * peak VO2 of less than or equal to 80% of predicted based on age and gender as determined by cardiopulmonary exercise testing

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for ≥7 days after stopping study drug
* Patients with a resting or provokable left ventricular outflow tract gradient of greater than or equal to 30mm Hg
* Septal reduction procedure within 3 months of the screening/baseline visit
* History of atrial fibrillation within 6 months of the screening/baseline visit or placement of ICD for secondary prevention
* Patients with a peak VO2 on the screening/baseline cardiopulmonary exercise test of > 80% of predicted based on age and gender
* Patients who require treatment with ACE inhibitors, angiotensin receptor blockers (ARBs), or renin inhibitors
* Known infiltrative or storage disorder such as Fabry disease, or amyloidosis
* Known or suspected symptomatic coronary artery diseases or evidence of prior myocardial infarction
* Systolic blood pressure of <100 mmHg or symptomatic hypotension during the screening/baseline period or treatment run-in period
* Contraindication to ARB administration or prior history of angioedema
* Persistent uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (5):
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Morristown, New Jersey
  - Novartis Investigative Site, Portland, Oregon
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion Crete
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Germany (4 sites), Greece (2 sites), Korea (2 sites), Spain (4 sites), United Kingdom (1 site), United States (5 sites)
Pre-assignment Details: Patients who met eligibility criteria entered a single-blind treatment run-in period. Patients who were unable to tolerate either placebo or the 50 mg p.o. b.i.d. dose level,were considered treatment run-in failures and were not randomized into the double-blind, placebo-controlled study
Groups:
- Run-in (All Participants): All patients received oral (p.o.) placebo b.i.d. for 2 weeks, followed by 50 mg p.o. b.i.d. of active LCZ696 for 2 weeks
Period: Treatment run-in Period
Arm/Group | Run-in (All Participants) | LCZ696 BID | Placebo BID
Started | 46 | 0 | 0
Completed | 40 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Screen Failure | 1 | 0 | 0
Period: Randomized Treatment Period
Arm/Group | Run-in (All Participants) | LCZ696 BID | Placebo BID
Started | 0 | 20 | 20
Randomized Analysis Set (The randomized analysis set (RAS) consisted of all randomized patients.) | 0 | 20 | 20
Per Protocol Analysis Set (The per-protocol analysis set (PPS) is a subset of the RAS that consists of all randomized patients who had no major protocol deviations with relevant impact on pharmacodynamics/efficacy data and who are at least 80% compliant with the overall study drug administration.) | 0 | 19 | 19
Completed | 0 | 17 | 19
Not Completed | 0 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-in (All Participants) | LCZ696 BID | Placebo BID | Total
Number analyzed (Participants) | 6 | 20 | 20 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (17.19) | 54.5 (11.84) | 57.2 (14.29) | 55.7 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 12
  Male | 3 | 17 | 14 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3 | 6
  White | 5 | 18 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak VO2 as Measured by Cardiopulmonary Exercise Test (CPET)
Description: The primary analysis assessed the effect of LCZ696 on the change from baseline in peak Volume of Oxygen (VO2) (ml/kg/min) at week 50 compared to placebo, where baseline peak VO2 came from the screening/baseline CPET.
  An increase in peak VO2 (mL/kg/min)/positive change is considered beneficial for the patient.
Time Frame: Baseline to 50 weeks
Population: Patients in the per protocol analysis set with and available value for the outcome measure at baseline and Week 50 .
  Per protocol analysis set consists of all randomized patients who had no major protocol deviations with relevant impact on PD/efficacy data and who are at least 80% compliant with the overall study drug administration.
Measure: Least Squares Mean (90% Confidence Interval); unit: mL/kg/min
Arm/Group | LCZ696 BID | Placebo BID
Number analyzed (Participants) | 18 | 19
mL/kg/min | 1.00 [-0.22 to 2.23] | 0.39 [-0.80 to 1.58]
Statistical Analysis 1: Comparison: LCZ696 BID vs Placebo BID; Test type: Superiority; p = 0.5506, longitudinal mixed effects (MMRM) model; Median Difference (Net) = 0.61, 80% CI 2-sided [-0.71 to 1.94]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 54 weeks.
Groups:
- Run-In Period Placebo: All patients received oral (p.o.) placebo b.i.d. for 2 weeks
- Run-In LCZ696 50 mg: All patients received 50 mg p.o. b.i.d. of active LCZ696 for 2 weeks
- Double-blind Period Placebo: Patients in the double-blind period treated with placebo
- Double-blind Period LCZ696 50 mg: Patients in the double-blind period treated with LCZ696 50mg
- Double-blind Period LCZ696 100 mg: Patients in the double-blind period treated with LCZ696 100mg
- Double-blind Period LCZ696 200 mg: Patients in the double-blind period treated with LCZ696 200mg
- Double-blind Period LCZ696: All patients in the double-blind period treated with LCZ696
- Total: Total
Arm/Group | Run-In Period Placebo | Run-In LCZ696 50 mg | Double-blind Period Placebo | Double-blind Period LCZ696 50 mg | Double-blind Period LCZ696 100 mg | Double-blind Period LCZ696 200 mg | Double-blind Period LCZ696 | Total
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/43 | 0/20 | 0/1 | 0/20 | 0/17 | 0/20 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/43 | 0/20 | 0/1 | 1/20 | 2/17 | 3/20 | 3/46
Other Adverse Events (participants affected / at risk) | 4/46 | 4/43 | 10/20 | 1/1 | 6/20 | 7/17 | 12/20 | 26/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period Placebo (N=46) | Run-In LCZ696 50 mg (N=43) | Double-blind Period Placebo (N=20) | Double-blind Period LCZ696 50 mg (N=1) | Double-blind Period LCZ696 100 mg (N=20) | Double-blind Period LCZ696 200 mg (N=17) | Double-blind Period LCZ696 (N=20) | Total (N=46)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.99% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period Placebo (N=46) | Run-In LCZ696 50 mg (N=43) | Double-blind Period Placebo (N=20) | Double-blind Period LCZ696 50 mg (N=1) | Double-blind Period LCZ696 100 mg (N=20) | Double-blind Period LCZ696 200 mg (N=17) | Double-blind Period LCZ696 (N=20) | Total (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 5
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 2 | 2 | 5
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04164732/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT04164732/SAP_001.pdf